CLINICAL TRIAL: NCT02516566
Title: Effects of Positive End-Expiratory Pressure Ventilation on Optic Nerve Sheath Diameter in Patients Undergoing Robot-Assisted Laparoscopic Prostatectomy
Brief Title: Effects of PEEP on Optic Nerve Sheath Diameter During Robot-Assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AsanMC
Record Dates: First submitted 2015-08-03; First posted 2015-08-06 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Other Surgical Procedures
Keywords: Positive end-expiratory pressure ventilation; Optic nerve sheath diameter

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEEP group (Experimental): Mechanical ventilation with PEEP 8 cmH2O
  Interventions: Other: PEEP
- No PEEP group (No Intervention): Mechanical ventilation with no PEEP

INTERVENTIONS:
Other: PEEP — Mechanical ventilation with PEEP 8 cmH2O
  Arms: PEEP group

SUMMARY:
The investigators aim to investigate the effects of positive end-expiratory pressure ventilation on intracranial pressure assessed by sonographic optic nerve sheath diameter in patients undergoing robot-assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
Effects of positive end-expiratory pressure ventilation on intracranial pressure have not been evaluated in patients undergoing laparoscopic surgery. We aim to investigate the effects of positive end-expiratory pressure ventilation on intracranial pressure assessed by sonographic optic nerve sheath diameter in patients undergoing robot-assisted laparoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo robot-assisted laparoscopic prostatectomy

Exclusion Criteria:

* Patients who have cerebrovascular disease or history of cerebrovascular disease
* Patients who are younger than 20 years

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | intraoperative

SECONDARY OUTCOMES:
Peak airway pressure | intraoperative
Arterial blood pressure | intraoperative
Heart rate | intraoperative
Arterial carbon dioxide tension | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center

REFERENCES:
- [Derived] Chin JH, Kim WJ, Lee J, Han YA, Lim J, Hwang JH, Cho SS, Kim YK. Effect of Positive End-Expiratory Pressure on the Sonographic Optic Nerve Sheath Diameter as a Surrogate for Intracranial Pressure during Robot-Assisted Laparoscopic Prostatectomy: A Randomized Controlled Trial. PLoS One. 2017 Jan 20;12(1):e0170369. doi: 10.1371/journal.pone.0170369. eCollection 2017. PMID 28107408